CLINICAL TRIAL: NCT04423926
Title: A Phase II, Prospective, Single-center Study of Lenalidomide in Combination With CHOP in Patients With Untreated PTCL
Brief Title: Lenalidomide in Combination With CHOP in Patients With Untreated PTCL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-SR-429
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: PTCL, NOS; AITL; ALK- ALCL; Phase III-IV ALK+ ALCL; EATL
Keywords: PTCL; lenalidomide; untreated; CHOP
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — Lenalidomide; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide+CHOP (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 10mg/d#15mg/d#20mg/d#25mg/d d1~d10# 21days a cycle
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2 d1
Drug: Doxorubicin — Doxorubicin 50 mg/m2 d1
Drug: Vincristine — Vincristine 1.4mg/m2 (maximum 2mg) d1
Drug: Prednisolone — Prednisolone 60mg/m2 d1-5

SUMMARY:
The prognosis of PTCL (except early stage ALK+ ALCL) is dismal. Previous study showed that single agent lenalidomide showed promising therapeutic activity in patients with relapsed or refractory PTCL. The investigators therefore design this phase II study to investigate the safety and efficacy of lenalidomide in combination with CHOP in patients with treatment-naive PTCL.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed PTCL, NOS, AITL, ALK- ALCL, phase III-IV ALK+ ALCL, EATL according to WHO 2016 criteria.
2. ECOG PS 0-2
3. Age 18-70 years old
4. Expected survival ≥ 12 weeks
5. A measurable or evaluable disease at the time of enrolment (diameter ≥1.5cm)
6. Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements.
7. Female subjects in childbearing age, their serum or urine pregnancy test must be negative. All patients must agree to take effective contraceptive measures during the trial measures

Exclusion Criteria:

1. Women who are pregnant or lactating. Patients have breeding intent in 12 months or cannot take effective contraceptive measures during the trial measures
2. Active hepatitis B or hepatitis C virus infection, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV infected persons
3. Patients known to have varicella or herpes zoster virus infection
4. Previous exposure to any anti-tumor therapy
5. Poor hepatic and/or renal function, defined as total bilirubin, ALT, AST, Cr more than two fold of upper normal level,Ccr# 50 mL/min unless these abnormalities were related to the lymphoma
6. History of DVT or PE within past 12 months
7. Poor bone-marrow reserve, defined as neutrophil count less than 1.5×109/L or platelet count less than 75×109/L, unless caused by bone marrow infiltration
8. New York Heart Association class III or IV cardiac failure; or Ejection fraction less than 50%;or history of following disease in past 6 months: acute coronary syndrome#acute heart failure#severe ventricular arrhythmia
9. CNS or meningeal involvement
10. Known sensitivity or allergy to investigational product
11. Major surgery within three weeks
12. Patients receiving organ transplantation
13. Patients with secondary tumour, excluding cured (5 years without relapse) in situ Non-melanoma skin cancer. superficial bladder cancer, in situ cervical cancer, Gastrointestinal intramucous carcinoma and breast cancer
14. Presence of Grade III nervous toxicity within past two weeks
15. Active and severe infectious diseases
16. Any potential drug abuse, medical, psychological or social conditions whichmay disturb this investigation and assessment
17. In any conditions which investigator considered ineligible for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2020-06-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose and dose limited toxicity | At the end of the first cycle of lenalidomide+CHOP (each cycle is 21 days)
Overall response rate | 6 months
  overall response rate after treated by lenalidomide-CHOP regimen

SECONDARY OUTCOMES:
Progressive free survival | 2 years
  from date of inclusion to date of progression, relapse, or death from any cause
Overall survival | 2 years
  from the date of inclusion to date of death, irrespective of cause

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, M.D., Ph.D., Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (1):
- The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hopfinger G, Nosslinger T, Lang A, Linkesch W, Melchardt T, Weiss L, Egle A, Greil R. Lenalidomide in combination with vorinostat and dexamethasone for the treatment of relapsed/refractory peripheral T cell lymphoma (PTCL): report of a phase I/II trial. Ann Hematol. 2014 Mar;93(3):459-62. doi: 10.1007/s00277-014-2009-0. Epub 2014 Jan 18. PMID 24441915
- [Background] Morschhauser F, Fitoussi O, Haioun C, Thieblemont C, Quach H, Delarue R, Glaisner S, Gabarre J, Bosly A, Lister J, Li J, Coiffier B. A phase 2, multicentre, single-arm, open-label study to evaluate the safety and efficacy of single-agent lenalidomide (Revlimid) in subjects with relapsed or refractory peripheral T-cell non-Hodgkin lymphoma: the EXPECT trial. Eur J Cancer. 2013 Sep;49(13):2869-76. doi: 10.1016/j.ejca.2013.04.029. Epub 2013 May 31. PMID 23731832
- [Background] Iqbal J, Wright G, Wang C, Rosenwald A, Gascoyne RD, Weisenburger DD, Greiner TC, Smith L, Guo S, Wilcox RA, Teh BT, Lim ST, Tan SY, Rimsza LM, Jaffe ES, Campo E, Martinez A, Delabie J, Braziel RM, Cook JR, Tubbs RR, Ott G, Geissinger E, Gaulard P, Piccaluga PP, Pileri SA, Au WY, Nakamura S, Seto M, Berger F, de Leval L, Connors JM, Armitage J, Vose J, Chan WC, Staudt LM; Lymphoma Leukemia Molecular Profiling Project and the International Peripheral T-cell Lymphoma Project. Gene expression signatures delineate biological and prognostic subgroups in peripheral T-cell lymphoma. Blood. 2014 May 8;123(19):2915-23. doi: 10.1182/blood-2013-11-536359. Epub 2014 Mar 14. PMID 24632715
- [Background] Schmitz N, de Leval L. How I manage peripheral T-cell lymphoma, not otherwise specified and angioimmunoblastic T-cell lymphoma: current practice and a glimpse into the future. Br J Haematol. 2017 Mar;176(6):851-866. doi: 10.1111/bjh.14473. Epub 2016 Dec 16. PMID 27982416